CLINICAL TRIAL: NCT02456883
Title: A Phase 1, Open-label Study to Investigate the Absorption, Metabolism and Excretion of [14C] ASP2215 in Patients With Advanced Solid Tumors
Brief Title: Study to Investigate the Absorption, Metabolism and Excretion of [14C] ASP2215 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0105
Expanded Access: NCT03070093 (Approved for marketing)
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors; Pharmacokinetics of 14C-labeled Gilteritinib
Keywords: ASP2215; 14C-labeled gilteritinib; Advanced Solid Tumors; Pharmacokinetics; gilteritinib
MeSH Terms: interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gilteritinib and 14C-labeled gilteritinib (Experimental): Gilteritinib will be taken once daily on study days 1 through 14 and days 16 through 47. On day 15, each participant will be given a single dose of 14C-labeled gilteritinib.
  Interventions: Drug: gilteritinib; Drug: 14C-labeled gilteritinib

INTERVENTIONS:
Drug: gilteritinib — oral
  Other Names: ASP2215
Drug: 14C-labeled gilteritinib — oral

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of 14C-labeled gilteritinib, in particular, the routes of excretion and extent of metabolism of gilteritinib following administration of a single dose of 14C-labeled gilteritinib after repeated doses of gilteritinib.

This study will also evaluate the safety of repeated oral administration of gilteritinib in subjects with advanced solid tumors as well as identify the metabolic profile of gilteritinib in plasma, urine and feces after a single oral dose of 14C-labeled gilteritinib.

DETAILED DESCRIPTION:
Participants will be admitted for evaluation to the clinical research unit on day 14 for potentially up to 14 days (day 29). At approximately days 36 and 45 participants will return to the clinic (for 3 days) for additional sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Subject had histologically or cytologically confirmed diagnosis of advanced solid tumor (measurable or nonmeasurable disease) for which no standard therapy is available.
* Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Subject must have a life expectancy > 12 weeks.
* Subject must have recovered from the effects of prior systemic antineoplastic or radiation therapy(s) to ≤ Grade 1 (National Cancer Institute - Common Terminology Criteria for Adverse Events [NCI-CTCAE], Version 4.0) severity or to subject's baseline values, excluding alopecia.
* Subject has adequate bone marrow, renal and hepatic function at baseline, as demonstrated by the following:

  * Absolute neutrophil count (ANC) ≥ 1500 cells/mm3
  * Platelet count ≥ 100,000 cells/mm3
  * Hemoglobin (Hb) ≥ 9 g/dL
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance > 60 mL/min if the serum creatinine is > 1.5 x ULN
  * Total bilirubin ≤ 1.5 x ULN
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 x ULN (or < 5 x ULN in subjects with liver metastases or hepatocellular carcinoma).
* Female subject must either:

  * Be of nonchildbearing potential: postmenopausal (defined as at least 1 year without any menses) prior to screening, or documented surgically sterile
  * Or, if of childbearing potential: agree not to try to become pregnant during the study and for 60 days after the final study drug administration and have a negative serum or urine pregnancy test at screening, and if heterosexually active, agree to consistently use 2 forms of birth control (at least one of which must be a barrier method) starting at screening and throughout the study period and for 60 days after final study drug administration.
* Female subject must not be breastfeeding at screening or during the study period, and for 60 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period and for 60 days after final study drug administration.
* Male subject and a female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (one of which must be a barrier method) starting at screening and continue throughout the study period and for 120 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 120 days after final study drug administration.
* Subject must be willing to comply with all procedures and assessments.

Exclusion Criteria:

* Subject has received more than 5 prior cytotoxic agent-containing regimens.
* Subject has symptomatic central nervous system (CNS) metastases or leptomeningeal involvement as assessed through medical history review and physical examination. Subject with prior brain metastases must:

  * have stable neurologic status post administration of local therapy (surgery or radiation) for a minimum of 2 weeks following completion of the definitive therapy.
  * be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events (AEs).
* Subject has had major surgery within 4 weeks prior to the first study dose.
* Subject has had chemotherapy within 4 weeks prior to the first study dose.
* Subject has had radiation therapy within 4 weeks prior to the first study dose.
* Subject with known hepatitis B surface antigen (HBsAg) positive status; or known or suspected active hepatitis C infection; or known human immunodeficiency virus (HIV) positive.
* Subject with malabsorption syndrome or disease or condition significantly affecting gastrointestinal function.
* Subject with significant or uncontrolled cardiac, renal, hepatic or other systemic disorders; or significant psychological conditions at baseline that in the investigator's opinion, makes the subject unsuitable for study participation.
* Subject with electrocardiogram (ECG) abnormalities on a 12-lead ECG performed within 14 days before start of the study drug that are considered by the Investigator to be clinically significant.
* Subject who has received strong or moderate inhibitors (e.g., ketoconazole or fluconazole) or inducers (e.g., rifampin or phenytoin) of cytochrome P450 (CYP)3A4 or of P-glycoprotein (P-gp), or substrates of multidrug and toxin extrusion (MATE)1 with the exception of antibiotics, antifungals, and antivirals that are used as standard of care post transplant or to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the subject within 2 weeks prior to start of study treatment and while on study.
* Subject requires treatment with concomitant drugs that target serotonin 5HT1R or 5HT2BR receptors or sigma nonspecific receptor, with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject has participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to the initiation of screening.
* Subject has a known history of serious hypersensitivity to ASP2215, or any component of the formulation used.
* Subject who has an ongoing toxicity ≥ Grade 2 (Common Terminology Criteria for Adverse Event [CTCAE] v4.03) attributable to prior medication to treat solid tumor (except alopecia) at the time of screening.
* Subject has had any of the following within 14 days prior to the first dose of study drug:

  * blood transfusion or hemopoietic factor therapy
  * evidence of active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity in whole blood): AUCtau | Days 15 - 46
  Area under the concentration curve over the dosing interval (AUCtau)
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity in whole blood): Cmax | Days 15 - 46
  Maximum concentration (Cmax)
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity in whole blood): tmax | Days 15 - 46
  Time of maximum concentration (tmax)
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity in whole blood): t1/2 | Days 15 - 46
  Terminal elimination half-life (t1/2)
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity in whole blood): CL/F | Days 15 - 46
  Apparent body clearance after extravascular dosing (CL/F)
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity in plasma): AUCtau | Days 15 - 46
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity in plasma): Cmax | Days 15 - 46
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity in plasma): tmax | Days 15 - 46
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity in plasma): t1/2 | Days 15 - 46
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity in plasma): CL/F | Days 15 - 46
Pharmacokinetics of 14C-labeled gilteritinib (Radioactivity ratio of whole blood/plasma concentrations): AUC | Days 15 - 46
  Area under the concentration (AUC)
Excretion rate of 14C-labeled gilteritinib (radioactivity in urine) | Days 15 - 46
  Percent of dose excreted in urine
Cumulative excretion of 14C-labeled gilteritinib (radioactivity in urine) | Days 15 - 46
  Cumulative total of radioactivity excreted in urine
Excretion rate of 14C-labeled gilteritinib (radioactivity in feces) | Days 15 - 46
  Percent of dose excreted in feces
Cumulative excretion of 14C-labeled gilteritinib (radioactivity in feces) | Days 15 - 46
  Cumulative total of radioactivity excreted in feces
Pharmacokinetics of gilteritinib (in plasma): AUCtau | Days 15 - 46
Pharmacokinetics of gilteritinib (in plasma): Cmax | Days 15 - 46
Pharmacokinetics of gilteritinib (in plasma): tmax | Days 15 - 46
Pharmacokinetics of gilteritinib (in plasma): CL/F | Days 15 - 46
Pharmacokinetics of gilteritinib (in urine): Aetau | Days 15 - 46
  Cumulative amount of study drug excreted into urine from the time of dosing to the start of the next dosing interval (Aetau)
Pharmacokinetics of gilteritinib (in urine): CLR | Days 15 - 46
  Renal clearance (CLR)
Pharmacokinetics of gilteritinib (in urine): AETAU% | Days 15 - 46
  Percentage of study drug dose excreted into urine over the time interval between consecutive dosing (AETAU%)

SECONDARY OUTCOMES:
Metabolite identification of gilteritinib in plasma, urine and feces | Days 15 - 46

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Site US10001, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] James AJ, Smith CC, Litzow M, Perl AE, Altman JK, Shepard D, Kadokura T, Souda K, Patton M, Lu Z, Liu C, Moy S, Levis MJ, Bahceci E. Pharmacokinetic Profile of Gilteritinib: A Novel FLT-3 Tyrosine Kinase Inhibitor. Clin Pharmacokinet. 2020 Oct;59(10):1273-1290. doi: 10.1007/s40262-020-00888-w. PMID 32304015
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=294